CLINICAL TRIAL: NCT01446770
Title: A Prospective, Randomized, Comparative Feasibility Study Evaluating the Initial Safety and Efficacy of Keloid Lesions Treated With MF-4181 Adjunctive to Surgical Scar Revision
Brief Title: Evaluation of the Initial Safety and Efficacy of Keloid Lesions Treated With MF-4181
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halscion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAL-0127
Record Dates: First submitted 2011-10-02; First posted 2011-10-05 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hydrogel scaffold (MF-4181) — Following surgical removal of the ear keloid, the incision will be treated with MF-4181.
  Other Names: Hydrogel scaffold

SUMMARY:
The objective of the study is to evaluate the initial safety and efficacy of MF-4181, a hydrogel scaffold, in the reduction of the volume, appearance, and/or symptoms associated with keloid scarring in subjects undergoing surgical revision of keloid scars.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 15 to 50 years of age each having at least one keloid scar on the ear. (If both ears have keloids, both ears may be treated with E-Matrix).
* Keloids that have not undergone more than two surgical revisions (laser, cryotherapy or surgery)
* Keloids that have been present for ≥ 1 year.
* The keloid must measure ≥ 0.5 cm and not extend onto other portions of the head, neck, or face.
* Able and willing to give written informed consent. (Age 15-17 must have written informed consent of legal guardian).
* Willing to comply with the follow up schedule for a minimum of 6 months.

Exclusion Criteria:

* Subjects with history of prior treatment at the study site or prior treatment of the keloid in the previous 6 weeks.
* Pregnant or planning to become pregnant during the course of the study.
* Heart disease or history of congestive heart failure.
* Advanced or poorly controlled diabetes.
* Current or history of heavy smoking (i.e., 10 pack years)
* Active local infection at the treatment site and/or systemic infection.
* History of or active central nervous system disease.
* History of fever, migraine headaches, and/or recurrent upper respiratory infection.
* Active collagen vascular disease or vasculitis, e.g., systemic lupus erythematosus, polyarthritis, dermatomyositis, systemic scleroderma or thrombotic thrombocytopenic purpura.
* Unwilling or unable to return for follow-up visits.
* Unwilling to refrain from use of any other scar treatment therapy/scar improving product, during the study, including steroid injections.
* Regular, continuous use of systemic corticosteroid therapy or topical corticosteroid use in the area to be treated.
* Current participation or participation within the last 3 months in the study of an investigational drug, device, or biologic.
* Unable or unwilling to follow post-operative instructions.
* Known hypersensitivity to MF-4181, collagen, dextran, or any of its constituent materials.
* Known hypersensitivities to animal-based products
* Previous participation in this study to avoid multiple enrollments of an individual subject.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Device safety | 6 months
  Device safety is defined as the incidence of device related adverse events.

SECONDARY OUTCOMES:
Device efficacy | 12 months
  Evaluations of cosmesis, induration, erythema and pigmentation will be evaluated by the investigator.
Device efficacy | 12 months
  Volume and linear measurements will be taken by the investigator
Device efficacy | 12 months
  Subject evaluation of cosmesis, pain, tenderness, itching and scar satisfaction will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Srikanth Garikaparthi, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Nassau, The Bahamas